CLINICAL TRIAL: NCT06018571
Title: Burden of Illness and Treatment Assessment of Patients With Dry Eye Disease: A Cross-Sectional Survey of Real-World Patients With Dry Eye Disease in the US
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLIF606A1US10
Record Dates: First submitted 2023-08-15; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study employed secondary database analysis of the Adelphi Dry Eye Disease (DED) Disease Specific Programme™ (DSP™), a templatized cross-sectional survey with retrospective data collection that is administered by Adelphi to a convenience sample of patients diagnosed with DED, and their consulting physicians in the United States. In addition to the survey data, the DED DSP also included recorded medical history data as reported by physicians (optometrists, ophthalmologists or refractive surgeons).

ELIGIBILITY:
Inclusion Criteria:

Main Sample:

* ≥ 18 years of age.
* Physician-confirmed DED diagnosis (at time of data collection).

Xiidra® Oversample:

* ≥ 18 years of age.
* Physician-confirmed DED diagnosis (at time of data collection).
* Have a current prescription for Xiidra® for their DED (at time of data collection).

Exclusion Criteria:

Main Sample:

• Involved in a DED clinical trial (at time of data collection).

Xiidra® Oversample:

* Involved in a DED clinical trial (at time of data collection).
* Included in the main sample previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 946 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Impact of Dry Eye on Everyday Life questionnaire© (IDEEL) mean scores | Up to approximately 18 months
  Mean IDEEL score on Symptom Bother dimension: score range 0-100, where higher scores indicate greater bother. Mean IDEEL scores on Daily Activities, Emotional Impact, and Work dimensions: score range 0-100, where higher scores indicate lesser impact.
Work Productivity and Activity Impairment© (WPAI) mean scores | Up to approximately 18 months
  A higher score on the WPAI indicates greater impairment and loss of productivity.
Frequency of consultations | Up to approximately 18 months
Frequency of DED-related hospitalizations | Up to approximately 18 months
Number of emergency room (ER)/intensive care unit (ICU) admittances | Up to approximately 18 months
Duration of ER/ICU admittances | Up to approximately 18 months
Number of evaluations/tests administered | Up to approximately 18 months
Frequency of evaluations/tests administered | Up to approximately 18 months

SECONDARY OUTCOMES:
Number of patients with reasons for consultation, per category | Up to approximately 18 months
Number of patients with current (at time of data capture) treatment regimen (prescribed, over-the-counter [OTC] treatments) | Up to approximately 18 months
Number of patients with reasons for not currently receiving any treatment for patient's DED (where appropriate), per category | Up to approximately 18 months
Number of patients with reasons for switching away from previous treatment line (where appropriate), per category | Up to approximately 18 months
Number of patients with "other than cure their DED, the most important benefit a drug treatment could provide," per category | Up to approximately 18 months
Impact of Dry Eye on Everyday Life Treatment Satisfaction module© (IDEEL-TS©) mean score | Up to approximately 18 months
  Score range 0-100, where a higher score indicates greater satisfaction.
Number of physicians assessing reasons for choice of current treatment line, per category | Up to approximately 18 months
Number of physicians assessing areas of improvement for current treatment line, per category | Up to approximately 18 months
Number of patients for whom cost/reimbursement was a driving factor in selection of current treatment | Up to approximately 18 months
Number of patients who were adherent to their current treatment plan, per category, as assessed by the physician | Up to approximately 18 months
Number of patients who were compliant to their current treatment plan, per category, as assessed by the physician | Up to approximately 18 months
Number of physicians assessing attributes associated with ideal medication, per category | Up to approximately 18 months
Number of physicians assessing attributes associated with currently prescribed medication, per category | Up to approximately 18 months
Number of physicians assessing influences on treatment decisions, per category | Up to approximately 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States